CLINICAL TRIAL: NCT06606093
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center, Phase 3 Clinical Trial and Open-label Extension Clinical Trial to Evaluate the Efficacy and Safety of DWP16001 in Type 2 Diabetic Nephropathy with Moderate Renal Impairment Patients (CKD Stage 3)
Brief Title: Evaluate the Efficacy and Safety of DWP16001 in Type 2 Diabetic Nephropathy with Moderate Renal Impairment Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP16001309
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetic Nephropathy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: DWP16001 Placebo
- Enavogliflozin 0.3 mg once daily (Experimental)
  Interventions: Drug: DWP16001 0.3mg

INTERVENTIONS:
Drug: DWP16001 Placebo — 1 tablet, Orally, Once daily single dose
  Arms: Placebo
Drug: DWP16001 0.3mg — 1 tablet, Orally, Once daily single dose
  Arms: Enavogliflozin 0.3 mg once daily

SUMMARY:
This study aims to evaluate the efficacy and safety of DWP16001 in type 2 diabetic nephropathy with moderate renal impairment patients (CKD stage 3)

DETAILED DESCRIPTION:
The drug in this study is called enavogliflozin. Enavogliflozin, as a once-daily oral therapy for type 2 diabetes. This study aiming to evaluate its efficacy in patients with type 2 diabetic nephropathy with moderate renal impairment patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 19 years or older as of the date of written consent.
2. Patients with type 2 diabetes who have been on up to 3 antidiabetic medications at a stable dosage and regimen for at least 8 weeks prior to the Pre-Baseline Visit (Visit 1-1). For insulin, a fluctuation of within 10% during the 8 weeks prior to the Pre-Baseline Visit (Visit 1-1) is allowed.
3. Patients with a BMI of 18 to 45 kg/m² at the Screening Visit (Visit 1).
4. Patients whose test results from the investigational site's laboratory at the Screening Visit (Visit 1) meet all of the following criteria:

   * HbA1c: 7.0% ≤ HbA1c ≤ 10.0%
   * eGFR: 30 ≤ eGFR < 60 ml/min/1.73 m² (using the CKD-EPI formula)
5. Patients who are willing to cooperate and participate in this clinical trial after understanding the explanation of the trial and who can voluntarily sign the informed consent form.
6. Patients whose central laboratory results from the sample collected at the Pre-Baseline Visit (Visit 1-1) show an eGFR of 30 ≤ eGFR < 60 ml/min/1.73 m² (using the CKD-EPI formula).
7. Patients whose central laboratory results from the sample collected at the Pre-Baseline Visit (Visit 1-1) show an HbA1c of 7.0% ≤ HbA1c ≤ 10.0%.
8. Patients with a medication compliance rate of 70-130% during the Run-in Period, as confirmed at the Baseline Visit (Visit 2).

Exclusion Criteria:

1. Individuals diagnosed with renal diseases other than diabetic chronic kidney disease
2. Patients with uncontrolled hypertension (SBP ≥ 180 mmHg or DBP ≥ 110 mmHg)
3. Individuals diagnosed with type 1 diabetes (insulin-dependent diabetes) or diabetic ketoacidosis
4. Individuals who are undergoing dialysis at the time of the Screening Visit (Visit 1) or have a history of renal transplantation or medically significant renal disease/surgery (e.g., renal vascular occlusive disease, nephrectomy)
5. Individuals who have received cytotoxic treatment, immunosuppressive therapy, or immunotherapy for renal disease within 6 months of the Baseline Visit (Visit 2)
6. Individuals diagnosed with or treated for any of the following diseases within 3 months of the Screening Visit (Visit 1), as determined by the investigator to be clinically significant:

   * Severe heart disease [heart failure (NYHA class III and IV), ischemic heart disease (angina, myocardial infarction), peripheral vascular disease, individuals who have undergone percutaneous transluminal coronary angioplasty or coronary artery bypass grafting]

     * NYHA class:
     * Class I: No limitation on physical activity; no symptoms during ordinary activities
     * Class II: Slight limitation on physical activity; no symptoms at rest, but symptoms occur during ordinary activities
     * Class III: Marked limitation on physical activity; no symptoms at rest, but symptoms occur with less than ordinary activities
     * Class IV: Symptoms present even at rest, and worsened by any physical activity
   * Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic or mitral valve stenosis
   * Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, arrhythmia
   * Transient ischemic attack
   * Severe cerebrovascular diseases (e.g., stroke, cerebral infarction, cerebral hemorrhage)
7. Individuals requiring treatment due to dehydration from continuous diarrhea or vomiting, or those at risk of fluid volume depletion
8. Individuals unable to take medications orally, or with major gastrointestinal diseases or surgeries (e.g., gastrectomy, gastrointestinal bypass) that may affect drug absorption, distribution, metabolism, or excretion
9. Individuals with positive results from the serology tests at the Screening Visit (Visit 1):

   * Positive for HIV
   * Positive for HBsAg with HBV DNA ≥ 2000 IU/mL
   * Positive for Anti-HCV
10. Individuals with severe liver dysfunction at the Screening Visit (Visit 1) as follows:

    * AST or ALT > 3 times the upper limit of normal
    * Total bilirubin > 2 times the upper limit of normal
11. Individuals with more than a 25% change in eGFR between the Screening Visit (Visit 1) and the Baseline Visit (Visit 2)
12. Individuals with clinically significant severe infections (e.g., those requiring continuous antibiotic or immunotherapy) or severe trauma, as determined by the investigator
13. Individuals with a past or present diagnosis of malignant tumors (participation allowed if cured or if there has been no recurrence in the past 5 years)
14. Individuals with a history of hypersensitivity to the active ingredient or components of the investigational drug
15. Individuals with a history of alcohol or drug abuse within 12 months of the Screening Visit (Visit 1)
16. Individuals taking ACE inhibitors, ARBs, or renin inhibitors (allowed if taken at a stable dose and regimen for more than 8 weeks prior to the Pre-Baseline Visit (Visit 1-1))
17. Individuals requiring continuous systemic corticosteroid treatment (use of topical corticosteroids for joint, nasal, ocular, or inhalation administration, or temporary systemic corticosteroid use for contrast agent allergies or adverse event treatment/prevention is allowed)
18. Women of childbearing potential who do not agree to use appropriate contraception* during the trial A. Women over 50 years of age who have been amenorrheic for at least 12 months after discontinuing exogenous hormone therapy B. Women with a history of irreversible surgical infertility (e.g., hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) (tubal ligation not allowed) C. Women under 50 years of age who have been amenorrheic for at least 12 months after discontinuing exogenous hormone therapy and whose luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within postmenopausal ranges according to the investigational site's standards Appropriate contraception: Complete abstinence, tubal ligation, hormonal contraceptives with no known drug interactions [levonorgestrel intrauterine system (IUS) (Mirena), medroxyprogesterone injection], copper intrauterine devices, and partner's vasectomy. Periodic abstinence (e.g., calendar methods, basal body temperature method, or post-ovulation method) and withdrawal are not considered acceptable contraceptive methods.
19. Men who have not undergone vasectomy and who do not agree to use barrier contraception (e.g., condoms), or whose partners do not agree to use appropriate contraception during the trial
20. Pregnant or breastfeeding women, or women with a positive pregnancy test result at the Screening Visit (Visit 1) or Baseline Visit (Visit 2)
21. Individuals who received investigational drugs within 8 weeks prior to the Screening Visit (Visit 1) (participation allowed if no investigational drug was administered or if involved in a non-interventional observational study)
22. Other individuals deemed inappropriate for trial participation at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c at Week 24 from Baseline after Randomization | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university ansan hospital, Ansan, Gyeongggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No